CLINICAL TRIAL: NCT03357107
Title: Evaluation of Local Control 2 Years After Robot-assisted Supraglottic Laryngectomy: a Multicenter Retrospective Study
Brief Title: Local Control After Robot-assisted Supraglottic Laryngectomy
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CRC_GHN_2017_009
Record Dates: First submitted 2017-11-23; First posted 2017-11-29 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Supraglottic Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Transoral robotic surgery (TORS) — All patients underwent primary tumour resection with transoral robotic surgery (TORS) using the daVinci robot (Intuitive Surgical, Sunnyvale CA)

SUMMARY:
Transoral robotic surgery is an option to treat supraglottic squamous cell carcinomas. Oncological outcomes 2 years after transoral robotic surgery for supraglottic laryngectomy were studied.

ELIGIBILITY:
Inclusion Criteria:

* Men or women over 18 years of age
* Patients with supra-glottic squamous cell carcinoma from T1 to T3, all stages N
* Patients with a robot assisted supra-glottic laryngectomy with at least 2 years follow-up

Exclusion Criteria:

* Patients for whom follow-up of at least 2 years has not been achieved;
* Major patients protected by the law (under guardianship or guardianship);
* Patients who expressed opposition to their participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with supraglottic squamous cell carcinoma who had undergone robot-assisted supraglottic laryngectomy and with at least 2 years follow-up
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Local control | 2 years after surgery
  Proportion of patients without cancer recurrence 2 years after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Croix-Rousse Hospital, Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No